CLINICAL TRIAL: NCT05813561
Title: A Multicenter, Randomized, Double-Blind, Active-Parallel-Controlled, Phase 3 Clinical Study to Investigate the Efficacy and Safety of DWP14012 in the Treatment of Reflux Esophagitis
Brief Title: The Efficacy and Safety of DWP14012 in Chinese Patients With Reflux Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP14012306
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — fexuprazan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP14012 (Experimental)
  Interventions: Drug: DWP14012
- Lansoprazole (Active Comparator)
  Interventions: Drug: DWP14012

INTERVENTIONS:
Drug: DWP14012 — DWP14012 40mg

SUMMARY:
To evaluate the efficacy, safety, and cost-effectiveness of DWP14012 40 mg compared to esomeprazole magnesium enteric-coated tablets for the treatment of reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for this study:

  1. Male or female subjects aged 18-75 years (inclusive);
  2. Subjects with a confirmed diagnosis of reflux esophagitis (Grade A-D according to LA classification) by esophagogastroduodenoscopy (EGD) at our site within 7 days prior to Visit 2 (date of randomization).
  3. Able to understand the information provided and to comply with protocol requirements;
  4. Voluntarily agreed to participate in this clinical study and signed the informed consent form (ICF).

Exclusion Criteria:

* 1）Subjects who were allergic to the investigational drug and any of its components or esomeprazole magnesium enteric-coated tablets, other benzimidazole compounds and their components; 2）Subjects who were unable to undergo esophagogastroduodenoscopy (EGD); 3）Subjects with eosinophilic esophagitis, Barrett's esophagus (≥ 3 cm), gastroesophageal varices, stricture of oesophagus, active peptic ulcer, active upper/lower gastrointestinal bleeding, or malignancies confirmed by EGD; 4）Subjects with Zollinger-Ellison syndrome, achalasia, irritable bowel syndrome, or inflammatory bowel disease; 5）Subjects with concomitant diseases that may affect esophageal motility (e.g., dermatosclerosis, viral infection or fungal infection, etc.), or a history of esophageal radiotherapy or esophageal cryotherapy; 6）Subjects who had undergone surgery to reduce gastric acid secretion, or any surgery that affected the structure or function of the esophagus, stomach, or duodenum (excluding benign tumor excision, endoscopic resection of benign polyps, and simple suture procedures such as gastric perforation); 7）Subjects with warning symptoms (e.g., odynophagia, severe dysphagia, bleeding, weight loss, anemia, or hematochezia) of gastrointestinal malignancies (excluding those who did not have any endoscopically confirmed anatomical abnormalities of the esophagus or stomach); 8）Subjects with a medical history of serious hepatic, renal, neurological, respiratory, endocrine, hematological, cardiovascular, or genitourinary diseases; 9）Subjects with a history of malignancies within 5 years prior to screening (excluding those who had recovered from non-digestive malignancies for 5 years and have not relapsed); 10）Subjects with a medical history of psychiatric disorders (excluding those with psychiatric disorders who were currently stable as judged by the investigator and were not receive treatment), or drug or alcohol abuse within 12 months prior to screening; 11）Subjects who required continuous treatment with nonsteroidal anti-inflammatory drugs (e.g., aspirin), systemic glucocorticoids, and antithrombotic drugs during the study (excluding those who used low-dose aspirin [≤ 100 mg/day] prophylactically); 12）Subjects who were taking anti-retroviral drugs such as atazanavir and nelfinavir at screening; 13）Subjects who used therapeutic doses of drugs for gastroesophageal reflux disease within 7 days prior to randomization, such as proton pump inhibitors, potassium competitive acid blockers, histamine H2 receptor antagonists, mucosal protective drugs, drugs promoting gastrointestinal motility, and traditional Chinese medicinal products for gastroesophageal reflux disease; 14）Subjects with alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin ≥ 2 × upper limit of normal (ULN); creatinine (Scr) ≥ 1.5 × ULN at screening; 15）Subjects who were positive for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg) and/or hepatitis C virus (HCV) antibodies at screening; 16）Pregnant or lactating women; subjects of childbearing potential who were unable or unwilling to use adequate contraception from the time of signing the ICF until 30 days after the last dose or their partners were unwilling to use contraception; 17）Subjects who have participated and received treatment in clinical studies of other drugs, devices, etc. within 3 months prior to screening; 18）Subjects who were ineligible (for any reason) to participate in the study as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
mucosal healing within 8 weeks | 8weeks
  The percentage of subjects with endoscopically confirmed mucosal healing within 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: The First Affiliated Hospital of Sun Yat-sen University Chen, M.D., Ph.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Minhu Chen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhuang Q, Liao A, He Q, Liu C, Zheng C, Li X, Liu Y, Wang B, Liu S, Zhang Y, Lin R, Chen H, Deng M, Tang Y, He C, Dai W, Tang H, Gong L, Li L, Xu B, Yang C, Zhou B, Su D, Guo Q, Li B, Zhou Y, Wang X, Fei S, Wu H, Wei S, Peng Z, Wang J, Li Y, Wang H, Deng T, Ding S, Li F, Chen M, Xiao Y. The efficacy and safety of fexuprazan in treating erosive esophagitis: a phase III, randomized, double-blind, multicenter study. J Gastroenterol Hepatol. 2024 Apr;39(4):658-666. doi: 10.1111/jgh.16471. Epub 2024 Jan 22. PMID 38251791